CLINICAL TRIAL: NCT00590395
Title: The Utility of FDG-PET and PET/CT in the Evaluation of Patients With Suspected Cholecystitis
Brief Title: FDG-PET/CT in the Evaluation of Patients With Suspected Cholecystitis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Alan D. Waxman, M.D. (Other)
Responsible Party: Sponsor-Investigator, Alan D. Waxman, M.D., Director, Imaging / Nuclear Medicine / Nuclear Cardiology, Cedars-Sinai Medical Center
Organization: Cedars-Sinai Medical Center (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: CSMC IRB Pro00007311; CSMC216788 (Other: Cedars-Sinai Medical Center)
Record Dates: First submitted 2007-12-26; First posted 2008-01-10 (Estimated); Results first posted 2019-10-17 (Actual); Last update posted 2019-12-10 (Actual); Status verified 2019-12

CONDITIONS: Cholecystitis
Keywords: Cholecystitis; FDG PET/CT; HIDA scan
MeSH Terms: conditions — Cholecystitis | interventions — Fluorodeoxyglucose F18

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- FDG-PET/CT to determine Cholecystitis (Experimental): 19 patients with suspected acute cholecystitis and a positive HIDA will be included in the study. This is purposely a highly selective population which most likely will have surgical proof of the findings. Subjects will receive an FDG PET/CT exam to determine the presence of gallbladder inflammation/infection(cholecystitis). Please note that 18FDG is an FDA approved radiopharmaceutical.
  Interventions: Drug: 18FDG (an FDA-approved radiopharmaceutical)

INTERVENTIONS:
Drug: 18FDG (an FDA-approved radiopharmaceutical) — Route: Intravenous, Dosage: 5-10mCi, frequency: Single Administration
  Other Names: 2-deoxy-2-[18F] fluoro-D-glucose (18FDG)

SUMMARY:
This is a pilot study to investigate the ability of fluorodeoxyglucose-positron emission tomography (FDG-PET) and Positron emission tomography-computed tomography (PET/CT) as a direct method of detecting infection and/or inflammation of the gallbladder.

DETAILED DESCRIPTION:
Hepatobiliary iminodiacetic acid (HIDA) scan scintigraphy is a nuclear medicine scan used to evaluate patients suspected of having acute cholecystitis (infection/inflammation of the gallbladder). Because it is an indirect test that looks for obstruction of the cystic duct structure, there are many causes for a false-positive HIDA study. There is a need for a more sensitive and specific test that can accurately assess gallbladder infection and/or inflammation.

The purpose of this study is to determine the effectiveness of fluorodeoxyglucose (FDG) as a direct means of detecting patients with acute cholecystitis. FDG is an imaging agent that has previously been shown to accumulate in areas of infection and/or inflammation. The location and intensity of FDG accumulation in the body can be detected with a camera system called a "positron emission tomography" (PET) camera. In theory, this test should be effective in detecting acute infection and/or inflammation of the gallbladder.

Consenting participants will receive injection of FDG one hour prior to the FDG-PET/CT examination. The participant will then be imaged using a PET/CT machine, which is a special camera system that is capable of performing both a PET and CT scan at the same time. A CT scan is an anatomical imaging test and, for this research study, will mainly be used to localize the area of 18FDG accumulation recorded by the PET scan. The examination will take approximately one hour.

ELIGIBILITY:
Inclusion Criteria:

* known or high suspicion of cholecystitis
* highly likely to undergo cholecystectomy
* positive HIDA study
* age >18 years old
* provide written informed consent

Exclusion Criteria:

* highly unlikely to proceed to surgery or biopsy
* received an investigational drug within the past 30 days
* pregnant or lactating
* decline to provide written informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2007-07; Primary Completion 2010-01 (Actual); Study Completion 2010-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Alan D. Waxman, M.D., Principal Investigator — Cedars-Sinai Medical Center
Locations (1):
- Cedars-Sinai Medical Center, S. Mark Taper Foundation Imaging Center, Los Angeles, California, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Patients With Suspected Acute Cholecystitis: 19 patients with suspected acute cholecystitis and a positive hepatobiliary iminodiacetic acid (HIDA) will be included in the study. This is purposely a highly selective population which most likely will have surgical proof of the findings. Subjects will receive an FDG (fluorodeoxyglucose) Positron Emission Tomography - Computed Tomography (PET/CT) exam to determine the presence of gallbladder inflammation/infection(cholecystitis). Please note that 18FDG is an FDA approved radiopharmaceutical.
  18FDG (an FDA-approved radiopharmaceutical): Route: Intravenous, Dosage: 5-10mCi, frequency: Single Administration
Period: Overall Study
Arm/Group | Patients With Suspected Acute Cholecystitis
Started | 19
Completed | 19
Not Completed | 0

BASELINE CHARACTERISTICS:
Groups:
- Patients With Suspected Acute Cholecystitis: 19 patients with suspected acute cholecystitis and a positive HIDA will be included in the study. This is purposely a highly selective population which most likely will have surgical proof of the findings. Subjects will receive an FDG PET/CT exam to determine the presence of gallbladder inflammation/infection(cholecystitis). Please note that 18FDG is an FDA approved radiopharmaceutical.
  18FDG (an FDA-approved radiopharmaceutical): Route: Intravenous, Dosage: 5-10mCi, frequency: Single Administration
Arm/Group | Patients With Suspected Acute Cholecystitis
Number analyzed (Participants) | 19
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 13
  >=65 years | 6
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7
  Male | 12
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United States | 19

OUTCOME MEASURES:

1. Primary Outcome: Sensitivity and Specificity of FDG PET/CT and Tc99mHIDA in the Evaluation of Subjects Suspected of Cholecystitis
Description: Percent of patients identified of having cholecystitis using FDG PET/CT compared to patients identified of having pathological diagnosis of cholecystitis (sensitivity) Percent of patients identified of not having cholecystitis using FDG PET/CT compared to patients identified of not having pathological diagnosis of cholecystitis (specificity)
  * number of false positives = number of patients incorrectly identified of having cholecystitis using FDG PET/CT compared to a negative pathological diagnosis.
  * number of false negatives = number of patients incorrectly identified of not having cholecystitis using FDG PET/CT compared to a positive pathological diagnosis.
  * number of true positives = number of patients correctly identified of having cholecystitis using FDG PET/CT compared to a positive pathological diagnosis.
  * number of true negatives = number of patients correctly identified of not having cholecystitis using FDG PET/CT compared to a negative pathological diagnosis.
Time Frame: 1-2 days through the post operative period
Population: All patients
Measure: Count of Participants; unit: Participants
Groups:
- Suspected Acute Cholecystitis: 19 patients with suspected acute cholecystitis and a positive HIDA will be included in the study. This is purposely a highly selective population which most likely will have surgical proof of the findings. Subjects will receive an FDG PET/CT exam to determine the presence of gallbladder inflammation/infection(cholecystitis). Please note that 18FDG is an FDA approved radiopharmaceutical.
  18FDG (an FDA-approved radiopharmaceutical): Route: Intravenous, Dosage: 5-10mCi, frequency: Single Administration
Arm/Group | Suspected Acute Cholecystitis
Number analyzed (Participants) | 19
Participants
  +PET/CT: number analyzed (Participants) | 10
  +PET/CT: +Path | 9
  +PET/CT: -Path | 0
  +PET/CT: N/A Path | 1
  -PET/CT: number analyzed (Participants) | 9
  -PET/CT: +Path | 1
  -PET/CT: -Path | 2
  -PET/CT: N/A Path | 6

ADVERSE EVENTS:
Arm/Group | Suspected Acute Cholecystitis
All-Cause Mortality (participants affected / at risk) | 0/19
Serious Adverse Events (participants affected / at risk) | 0/19
Other Adverse Events (participants affected / at risk) | 0/19

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No